CLINICAL TRIAL: NCT04947748
Title: Short Post-operative Antibacterial Therapy in Complicated Appendicitis: Oral Versus Intravenous
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Estonia Medical Centre (Other)
Collaborators: Tartu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Acute Appendicitis; Acute Appendicitis With Rupture; Acute Appendicitis Without Peritonitis; Acute Appendicitis With Appendix Abscess; Appendicitis; Perforation; Appendicitis Perforated; Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24 hour intravenous antibacterial therapy (Active Comparator): S.Augmentin 1,2g x 3 i/v
  Interventions: Other: Oral versus intravenous administration of antibacterial treatment
- 24 hour oral antibacterial therapy (Experimental): T.Augmentin 1g x 3 p/o
  Interventions: Other: Oral versus intravenous administration of antibacterial treatment

INTERVENTIONS:
Other: Oral versus intravenous administration of antibacterial treatment — Mode of administration of antibacterial treatment

SUMMARY:
Short Post-operative Antibacterial Therapy in Complicated Appendicitis: Oral Versus Intravenous is a prospective randomized controlled trial comparing 24 hour intravenous antibacterial therapy to 24 hour oral antibacterial therapy after surgery in complicated appendicitis.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with acute appendicitis and are candidates for laparoscopic appendectomy.

Exclusion Criteria:

Patients with compromised immune system (HIV, diabetes), ongoing or completed radio-chemotherapy in past 5 years, prosthetic heart valve, vascular prosthesis, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Infectious complications | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Lipping, MD, Principal Investigator — North Estonia Medical Centre
Locations (1):
- North Estonia Medical Centre, Tallinn, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lipping E, Saar S, Reinsoo A, Bahhir A, Kirsimagi U, Lepner U, Talving P. Short Postoperative Intravenous Versus Oral Antibacterial Therapy in Complicated Acute Appendicitis: A Pilot Noninferiority Randomized Trial. Ann Surg. 2024 Feb 1;279(2):191-195. doi: 10.1097/SLA.0000000000006103. Epub 2023 Sep 25. PMID 37747168